CLINICAL TRIAL: NCT02322736
Title: A Prospective Observational Study of 1st and 2nd Line Vectibix® Use in KRAS/NRAS-wt mCRC Patients to Evaluate Pattern of Use and Overall Response Rates
Brief Title: Prospective Observational Study of 1st and 2nd Line Vectibix® Use in RAS-wt mCRC Pts to Evaluate Pattern of Use and ORR
Acronym: VISION
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: ZeinCRO Hellas SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120286
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer, wild type RAS, Panitumumab, Vectibix, Greece
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WT RAS mCRC: Wild Type RAS metastatic colorectal cancer patients

SUMMARY:
The study will shed additional light on the impact of Vectibix® under the current, standard clinical conditions of mCRC treatment in Greece. It will provide data on the duration and the outcomes of Vectibix® treatment in real-life setting.

DETAILED DESCRIPTION:
This is a single-arm, multi-center, prospective, observational, descriptive, noninterventional study in patients with mCRC in Greece who receive Vectibix®in 1st or 2nd line according to approved indication. The aim of the study is to obtain a clear understanding of the current practices concerning real-life treatment of mCRC patients with Vectibix® in first-line in combination with chemotherapy or second-line in combination with chemotherapy in Greece. This setting will also provide the opportunity to observe in a non-selected patient population with RAS WT mCRC the real-life habits of mCRC treatment, and in particular the duration and the outcomes of Vectibix® treatment. The data generated by this study may be used for reimbursement purposes, as it becomes an increasingly common need in Greece to provide locally generated data for use of drugs in the real-life setting to regulatory agencies and/or payors. Furthermore, this study could address the existing data gap in the treatment of anti-EGFR therapy beyond progression in the real-life setting.

Primary Objective(s): To describe the pattern of use of Vectibix® in combination with chemotherapy in 1st line or in 2nd line mCRC treatments as per approved Vectibix® indication.

Secondary Objective(s): To investigate the rate of objective response (ORR, defined as either a Complete Response or a Partial Response) and the rate of stable disease as best response in 1st line or in 2nd line chemotherapy regimens of mCRC including Vectibix®.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥18 years) at enrollment
* Histological documentation of mCRC diagnosis
* RAS WT tumor documented before study enrolment as per routine laboratory finding
* Subjects whose care will be managed primarily by the enrolling physician and/or all records will be available
* Measurable disease at baseline (preferably according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) if routinely used)
* Currently under (begin up to 8 weeks before informed consent) a 1st or 2nd line treatment regimen, including Vectibix® as per indication
* Tumor assessment (i.e. CT/MRI) within 16 weeks prior to first Vectibix® infusion
* Signed informed consent

Exclusion Criteria:

* Participation in any interventional clinical study (currently or during the three previous months from enrollment).
* Compromised ability to give informed consent (defined per clinical judgment).
* Unknown or mutant RAS tumor type

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target population will be adult patients (aged ≥ 18 years at enrollment) with a documented diagnosis of a RAS WT mCRC preferably measurable disease per modified Response Evaluation Criteria in Solid Tumors (RECIST v1.1) if routinely used, who are currently under (begin up to 8 weeks before informed consent) a 1st or 2nd line treatment regimen including Vectibix® as per indication.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
To describe the pattern of use of Vectibix® in combination with chemotherapy in 1st line or in 2nd line mCRC treatments as per approved Vectibix® indication. | 42 months
  Treatment patterns of Vectibix® and concomitant chemotherapy for mCRC will be decribed according to the following information:
  * Type of chemotherapy combined with Vectibix®
  * Starting dose and dose administration schedule of Vectibix® and chemotherapy
  * Cumulative dose, maximum dose, duration of exposure and total number of infusions received from the initiation of Vectibix® therapy and chemotherapy
  * Dose alterations for Vectibix and chemotherapy (including changes in frequency, reductions and/or delays).

SECONDARY OUTCOMES:
To investigate the rate of objective response (ORR, defined as either a Complete Response or a Partial Response) and the rate of stable disease as best response in 1st line or in 2nd line chemotherapy regimens of mCRC including Vectibix®. | 42 months
  Objective response rate (ORR) of the 1st line chemotherapy treatment including Vectibix®.
  Objective response rate (ORR) of the 2nd line chemotherapy treatment including Vectibix®.
  Stable disease rate (SD) of the 1st line chemotherapy treatment including Vectibix®.
  Stable disease rate (SD) of the 2nd line chemotherapy treatment including Vectibix®.

OTHER OUTCOMES:
Frequency of primary tumor resection, of metastatic lesion resection, of BRAF testing in the entire number of the study participants and frequency of BRAF mutation in the unselected Greek patient population with WT RAS mCRC included in the study. | 42 months
  Frequency of primary tumor resection in the entire number of the study participants (patients with WT RAS mCRC included in the study).
  Frequency of metastatic lesion resection in entire number of the study participants.
  Frequency of BRAF testing in the entire number of the study participants. Frequency of BRAF mutation in the unselected Greek patient population with WT RAS mCRC included in the study.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- Greece (11):
  - Research Site, Ampelokipoi, Athens
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Heraklion - Crete
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Maroussi, Athens
  - Research Site, Nea Kifissia, Athens
  - Research Site, Papagou
  - Research Site, Piraeus
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com